CLINICAL TRIAL: NCT05003765
Title: Are Superficial Parasternal Intercostal Plane (SPIP) Blocks With Local Anesthetic Alone and Local Anesthetic With Adjuvants Helpful in Managing Post-operative Pain in Coronary Artery Bypass Grafting (CABG)?
Brief Title: Are Superficial Parasternal Intercostal Plane (SPIP) Blocks With Bupivacaine and With or Without Adjuvants Helpful for Post-operative Pain After Coronary Artery Bypass Grafting?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Sandeep Krishnan, Clinical Associate Professor of Anesthesiology, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SPIP_Block
Record Dates: First submitted 2021-07-29; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Post-operative Pain Management
Keywords: coronary artery bypass grafting, superficial parasternal intercostal plane block , opioid consumption, magnesium, buprenorphine
MeSH Terms: interventions — Bupivacaine; Magnesium Sulfate; Buprenorphine

STUDY DESIGN:
Intervention Model Description: This study will consist of 4 arms (groups):
  Control Group (CTRL): No Block (Saline) Treatment Group1 (TRT1): SPIP Block with bupivacaine Treatment Group 2 (TRT2): SPIP Block with Bupivacaine +Magnesium as Adjuvant Treatment Group 3 (TRT3): SPIP Block with Bupivacaine +Magnesium + Buprenorphine both as Adjuvant
  Patients are assigned randomly to each group.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Saline injection (CTRL) (No Intervention): Arm 1- 50 Patients-Control Group (CTRL): No Block (Saline) Post-operatively patients will receive 20 mL of Saline (on each side) between the pectoralis major and external intercostal muscle aponeurosis at 2 cm lateral to the right and left of the sternal edge, corresponding to the fifth rib.
- SPIP Block (Experimental): Arm 2-50 Patients-Post-operatively patients will receive bilateral SPIP blocks by injecting 20 mL of 0.25% bupivacaine (on each side) between the pectoralis major and external intercostal muscle aponeurosis at 2 cm lateral to the right and left of the sternal edge, corresponding to the fifth rib.
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution
- SPIP Block + Magnesium (Experimental): Arm 3-50 Patients-Post-operatively patients will receive bilateral SPIP blocks by injecting 20 mL of 0.25% bupivacaine + 200mg of magnesium sulfate (on each side) between the pectoralis major and external intercostal muscle aponeurosis at 2 cm lateral to the right and left of the sternal edge, corresponding to the fifth rib.
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution, Magnesium Sulfate 200 mg
- SPIP Block + Magnesium + Buprenorphine (Experimental): Arm 4-50 Patients-Post-operatively patients will receive bilateral SPIP blocks by injecting 20 mL of 0.25% bupivacaine+ 200mg of magnesium sulfate + buprenorphine (300mcg) (on each side) between the pectoralis major and external intercostal muscle aponeurosis at 2 cm lateral to the right and left of the sternal edge, corresponding to the fifth rib.
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution, Magnesium Sulfate 200 mg, Buprenorphine 300 mcg

INTERVENTIONS:
Drug: Bupivacaine 0.25% Injectable Solution — Injection of Bupivacaine 0.25% Injectable Solution for SPIP Nerve Block.
  Arms: SPIP Block
Drug: Bupivacaine 0.25% Injectable Solution, Magnesium Sulfate 200 mg — Injection of Bupivacaine 0.25% Injectable Solution for SPIP Nerve Block. Addition of 200mg of magnesium sulfate as adjuvant.
  Arms: SPIP Block + Magnesium
Drug: Bupivacaine 0.25% Injectable Solution, Magnesium Sulfate 200 mg, Buprenorphine 300 mcg — Injection of Bupivacaine 0.25% Injectable Solution for SPIP Nerve Block. Addition of 200mg of magnesium sulfate and 300 mcg buprenorphine as adjuvants.
  Arms: SPIP Block + Magnesium + Buprenorphine

SUMMARY:
The purpose of this study is to determine whether the addition of the superficial parasternal intercostal plane (SPIP) block alone (30cc of 0.25% bupivacaine) or plus Magnesium (200mg of magnesium sulfate) or plus Magnesium + Buprenorphine (300mcg) as adjuvants can improve post-operative pain in patients undergoing cardiothoracic surgery, specifically, coronary artery bypass grafting (CABG)

DETAILED DESCRIPTION:
Postoperative pain management remains an important clinical challenge in cardiothoracic surgery. Inadequate postoperative pain control can have adverse pathophysiologic consequences, including increased myocardial oxygen demand, hypoventilation, suboptimal clearance of pulmonary secretions, acute respiratory failure, and decreased mobility, with associated increased risks for formation of clots in a blood vessels (thromboembolism). These adverse events may result in greater perioperative morbidity and mortality. Despite several multimodal approaches to postoperative pain control, optimal pain management after cardiothoracic procedures remains an issue.

Regional anesthesia is used to block sensation in a specific part of body during and after surgery. It offers numerous advantages over conventional general anesthesia, including faster recovery time, fewer side effects, no need for an airway device during surgery, and a dramatic reduction in post-surgical pain and reduction in opioid use following surgery. The use of local anesthetic peripheral nerve blocks for surgical anesthesia and postoperative pain management has increased significantly with the advent of ultrasound-guided techniques.

Ultrasound has revolutionized regional anesthesia by allowing real-time visualization of anatomical structures, needle advancement and local anesthetic (LA) spread. This has led not only to refinement of existing techniques, but also the introduction of new ones.

In particular, ultrasound has been critical in the development of fascial plane blocks, in which local anesthetic (LA) is injected into a tissue plane rather than directly around nerves. These blocks are believed to work via passive spread of LA to nerves traveling within that tissue plane, or to adjacent tissue compartments containing nerves.

Although research into these techniques is still at an early stage, the available evidence indicates that they are effective in reducing opioid requirements and improving the pain experience in a wide range of clinical settings. They are best employed as part of multimodal analgesia with other systemic analgesics, rather than as sole anesthetic techniques. Catheters may be beneficial in situations where moderate-severe pain is expected for >12 hours, although the optimal dosing regimen requires further investigation.

In this study the investigators will focus on the superficial parasternal-intercostal plane (SPIP) block, which is among the anteromedial chest wall (near sternum) blocks and was first performed by Raza et al. and Ohgoshi et al.

The investigators will be assessing whether the addition of SPIP block (alone or plus adjuvants) will decrease the visual analog scale (VAS) pain scores in the first 24 hours after surgery, decrease post-operative total opioid consumption (oral morphine equivalents), decrease total acetaminophen and ketorolac consumption, decrease post-operative nausea and vomiting (PONV), decrease length of the ICU stay, decrease time to extubation, and decrease length of hospital stay in comparison to when SPIP block is not administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary coronary artery bypass grafting

Exclusion Criteria:

* Patients with significant genetic or acquired clotting/bleeding disorders (hemophilia, DIC, etc.)
* Patients with significant platelet dysfunction
* Infection at site for regional anesthesia
* Allergy to local anesthetics
* Severe aortic stenosis
* Severe mitral stenosis
* Sepsis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative total opioid consumption (oral morphine equivalents) | 24 hours after the surgery
  Total Opioid consumption 24 hours post surgery oral moral morphine equivalents
Visual analog scale (VAS) pain scores | 6 hours after surgery
  Pain Scores measured via a Visual Analog Scale (0-10, Higher scores mean worse outcome)
Visual analog scale (VAS) pain scores | 12 hours after surgery
  Pain Scores measured via a Visual Analog Scale (0-10, Higher scores mean worse outcome)
Visual analog pain (VAS) scores | 24 hours after surgery
  Pain Scores measured via a Visual Analog Scale (0-10, Higher scores mean worse outcome)
Length of hospital stay (LOS) | Up to 1 month
  The days spent in the hospital from surgery to discharge

SECONDARY OUTCOMES:
Incidence of post-operation nausea and vomiting (PONV) | 24 hours
  The percentage of the patients who had post-operative nausea and vomiting (PONV) within 24 hours of surgery
Acetaminophen consumption | 24 hours
  Total acetaminophen consumption in mg 24 hr after surgery
NSAID (ketorolac) consumption | 24 hours after surgery
  Total NSAID consumption in mg
Length of ICU stay | Up to 1 month
  Length of stay in Intensive Care Unit from surgery to discharge from Intensive Care Unit
Time to extubation | 24 Hours
  Time it took for patient to be extubated

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph Mercy Oakland Hospital, Pontiac, Michigan, United States

IPD SHARING:
Plan to Share IPD: No